CLINICAL TRIAL: NCT01612169
Title: NIDA CTN Protocol 0049. Project HOPE -- Hospital Visit as Opportunity for Prevention and Engagement for HIV-Infected Drug Users
Brief Title: Hospital Visit as Opportunity for Prevention and Engagement for HIV-Infected Drug Users
Acronym: CTN0049
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Jackson Health System (Other); Grady Health System (Other); Johns Hopkins University (Other); Boston Medical Center (Other); Hahnemann University Hospital (Other); Rush University Medical Center (Other); PARKLAND HEALTH AND HUMAN SERVICES (Unknown); University of Pittsburgh (Other); University of California, Los Angeles (Other); University of Alabama at Birmingham (Other); St. Luke's-Roosevelt Hospital Center (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lisa Metsch, Stephen Smith Professor and Chair of the Department of Sociomedical Sciences, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAK1709; U10DA013720-11 (NIH)
Record Dates: First submitted 2012-06-04; First posted 2012-06-05 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: HIV; AIDS; Substance Abuse; Inpatient
Keywords: HIV patients; Hospitalized patients; Substance Users; Drug Users
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders; Drug Misuse | interventions — Patient Navigation; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment as Usual (TAU) Group (No Intervention): Participants assigned to the TAU group will receive the standard treatment provided at each hospital for linking patients to HIV and substance use care.
  During the formal site selection process, a thorough assessment will be conducted of each site's standard practice for linkage to HIV care and substance use treatment. Throughout the course of the trial, hospital sites will be monitored for any potential changes that might occur in standard practice around linkage to HIV care and substance use treatment.
- Patient Navigation (PN) Group (Experimental): The patient navigator approach includes five functions: 1) establishing an effective working relationship; 2) encouraging identification and use of strengths, abilities and assets; 3) supporting client control over goal setting and the search for needed resources; 4) viewing the community as a resource and identifying informal sources of support; and 5) conducting case management as an active community based activity.
  After the initial four meetings, patient navigators will meet with PN group participants ideally twice monthly during months 2 and 3 and once monthly during months 4 - 6.
  Interventions: Behavioral: Patient Navigation (PN) Group
- Patient Navigator Plus Contingency Management (PN+CM) Group (Experimental): Study participants randomized to this group will receive the patient navigation (PN) intervention as outlined above combined with contingency management (CM). Using the principles of contingency management, this combined intervention will incorporate viral load suppression as a target of reinforcement as well as several other behaviors (HIV clinical care, medication adherence, cessation or reduction of substance use) that are hypothesized to be moderators or mediators of the primary outcome.
  For participants randomly assigned to the PN+CM study group, patient navigators will: 1) effectively communicate the incentive plan to the participant, 2) track each of the seven target behaviors that may earn participant incentives, 3) verify occurrence of the target behaviors, 4) deliver incentives according to the protocol, and 5) maintain a record of incentives delivered. PNs will use a computer-based tracking program to facilitate this work.
  Interventions: Behavioral: Patient Navigator Plus Contingency Management (PN+CM) Group

INTERVENTIONS:
Behavioral: Patient Navigation (PN) Group — The patient navigator approach includes five functions: 1) establishing an effective working relationship; 2) encouraging identification and use of strengths, abilities and assets; 3) supporting client control over goal setting and the search for needed resources; 4) viewing the community as a resource and identifying informal sources of support; and 5) conducting case management as an active community based activity.
  Arms: Patient Navigation (PN) Group
Behavioral: Patient Navigator Plus Contingency Management (PN+CM) Group — Study participants randomized to this group will receive the patient navigation (PN) intervention as outlined above combined with contingency management (CM).
  Arms: Patient Navigator Plus Contingency Management (PN+CM) Group

SUMMARY:
Primary Objective: This study will evaluate the most effective strategy in achieving HIV virologic suppression among HIV-infected substance users recruited from the hospital setting who are randomly assigned to one of three treatment conditions: 1) Patient Navigator (PN); 2) Patient Navigator + Contingency Management (PN+CM); and 3) Treatment as Usual (TAU).

Primary Hypothesis: The rate of viral suppression (plasma HIV viral load of <= 200 copies/mL) relative to non-suppression or all-cause mortality in the 3 study groups will differ from each other at the 12 month follow-up.

Sub-hypothesis 1. The rate of virologic suppression (plasma HIV viral load of <= 200 copies/mL) in the PN+CM group will be greater than that in the TAU group.

Sub-hypothesis 2. The rate of virologic suppression in the PN+CM group will be greater than that in the PN group.

Sub-hypothesis 3. The rate of virologic suppression in the PN group will be greater than that in the TAU group.

Secondary Objectives:

1. To evaluate the effect of the experimental interventions on: HIV virological suppression and CD4 T-cell count changes at 6 months post-randomization; engagement in HIV primary care and visit attendance; and rate of hospitalizations.
2. To evaluate the effect of the experimental interventions on: drug use frequency and severity; and drug use treatment engagement and session attendance.
3. To assess selected mechanisms of action of the intervention (.i.e. mediators of intervention effect).
4. To assess potential characteristics associated with differential treatment effectiveness (i.e. moderators of intervention effect).
5. To evaluate the incremental cost and cost-effectiveness of the interventions.

DETAILED DESCRIPTION:
This study is a 3-arm randomized, prospective trial in which HIV-infected inpatients who report substance use at screening will be randomized in 1:1:1 ratio to Patient Navigator (PN) vs. Patient Navigator + Contingency Management (PN+CM) vs. Treatment as Usual (TAU). Randomization will occur after screening, informed consent, baseline assessment and collection of biological (blood) specimens. Participants assigned to the PN and PN+CM groups will meet (ideally at bedside if the participant is still hospitalized at the time of randomization) with the Patient Navigator interventionist and will complete up to 11 intervention sessions over the 6-month-long intervention period. Participants assigned to the TAU group will receive care as it is typically offered in the inpatient setting. Follow-up visits will be conducted at approximately 6 and 12 months post-randomization.

To minimize patient and staff burden, sites may implement a pre-screening procedure with permission from their respective IRBs to determine which inpatients would meet the study's AIDS-defining illness/CD4 count/viral load inclusion criteria. Pre-screening, screening, enrollment, assessment, randomization and the initial intervention visit will (ideally) occur during the participant's stay at an inpatient facility. Recognizing that participants may be recruited at various stages of illness during their inpatient visit, however, this may not be possible. To allow maximum flexibility, all activities that occur after the screening informed consent may be completed after the patient has been discharged from the hospital. The intervention duration will be 6 months with sessions ideally occurring weekly during the first month, bi-weekly during months 2 and 3 and monthly during months 4- 6. Follow-up visits will occur at approximately 6 and 12 months post-randomization. Therefore, the total duration of individual participation in the study is approximately 12 months.

Prior to approaching patients to recruit them into the study, members of the medical teams within each hospital (i.e., attending physicians, fellows, residents and nurse practitioners) who are involved in patient care and who know the patients' HIV-infected status will assess the medical stability of the patients. If a patient has expressed interest in potentially participating in research and is deemed medically stable, then a study staff member will meet with the patient at bedside to discuss the study. Strict ethical guidelines regarding professional conduct and confidentiality will be enforced for all study staff.

Prior to screening individuals to determine their eligibility to participate, the research staff will briefly explain the study purpose, procedures, potential risks and benefits and voluntary nature of participation. Individuals willing to be screened to determine eligibility will provide written informed consent, including providing HIPAA authorization for medical record abstraction. After signing the consent and HIPAA forms, participants will be offered copies of the forms to keep for their records.

After the enrollment process (providing written informed consent and completing a locator form) is complete and a brief rapport-building discussion between the interviewer and participant has taken place, the research interviewer will administer the baseline assessment through a handheld Computer Assisted Personal Interview (CAPI) device. The CAPI system displays each assessment question on a computer monitor, allowing the interviewer to read the questions and then enter the participants' responses directly into the computer. The baseline assessment will include, but not be limited to questions on participant demographics, HIV care, medication adherence, substance use and co morbid conditions such as hepatitis, depression, etc.

Collection of Biologic Specimens:

We will collect blood specimens at the baseline, 6-month and 12-month follow-up visits to evaluate the primary outcome, HIV virologic suppression, as well as to measure CD4 count, and complete blood count (CBC). Blood specimen processing will be done by sites' local laboratories. In the event that a blood specimen cannot be collected for any reason (e.g., vein is "dry", participant is lost to follow-up, etc.) or the result of a collected specimen is not available (e.g., not enough specimen drawn, lab processing error, etc.), the study team may abstract and use non-study lab results for the purpose of evaluating the HIV virologic suppression outcome and measuring CD4 count and CBC. Participants randomized to the intervention groups may also provide urine for drug screening.

Randomization:

Participants will be randomized in a 1:1:1 fashion to one of the 3 treatment groups. Randomization will be stratified by site. The randomization procedure will be conducted in a centralized process through the Data and Statistical Center (DSC2). After the baseline assessment is successfully completed, a designated study staff member will perform the randomization. Randomization for each participant is done over the Internet using the Enrollment Module in AdvantageEDC (the study electronic data capture system).

Study Interventions:

The 3 treatment conditions/study groups are: 1) Patient Navigator intervention (PN), 2) Patient Navigator plus Contingency Management (PN+CM) intervention and 3) Treatment as Usual (TAU).

The patient navigator (PN) approach includes five functions: 1) establishing an effective working relationship; 2) encouraging identification and use of strengths, abilities and assets; 3) supporting client control over goal setting and the search for needed resources; 4) viewing the community as a resource and identifying informal sources of support; and 5) conducting case management as an active community based activity. Specifically, patient navigators will provide the following to all study participants randomized to the PN group: 1) four initial meetings, ideally having the first one during hospitalization and three within the first 3 weeks of hospital discharge, and 2) after the initial four meetings, patient navigators will meet with the PN group participants ideally twice monthly during months 2 and 3 and once during months 4 - 6.

Study participants randomized to the patient navigator plus contingency management (PN+CM) group will receive the patient navigation (PN) intervention as outlined above and in Section 11.2 of the sponsor protocol combine with contingency management (CM). For participants randomly assigned to the PN+CM study group, patient navigators will: 1) effectively communicate the incentive plan to the participant, 2) track each of the seven target behaviors that may earn participant incentives, 3) verify occurrence of the target behaviors, 4) deliver incentives according to the protocol, and 5) maintain a record of incentives delivered.

Participants assigned to the treatment as usual (TAU) group will receive the standard treatment provided at participating sites for linking patients to HIV and substance use care.

Follow-up visits will be conducted at approximately 6- and 12-months post-randomization and will involve follow-up CAPIs and blood collection.

ELIGIBILITY:
Inclusion Criteria

Participating individuals must:

1. be admitted to a hospital and be HIV-infected at the time of recruitment
2. be at least 18 years old
3. meet one of the following: A) have an AIDS-defining illness during the current hospital admission; or B) have the most recent CD4 count and viral load performed within the past 6 months be <350 cells/uL and >200 copies/mL; or C) have the most recent CD4 count and viral load performed within the past 12 months be <=500 cells/uL and >200 copies/mL or unknown accompanied by the Site PI's discretion that the patient a) is likely to currently have a viral load >200 copies/mL, b) is not currently successfully/correctly taking antiretroviral therapy (ART) and c) needs to be on ART
4. report (or have evidence in the medical record of) any opioid and/or stimulant and/or heavy alcohol use within the past 12 months (Note: Medical record evidence may consist of a) positive toxicology screen(s) for stimulants or heavy alcohol or b) clinician notes indicating heavy use of alcohol, use of stimulants or non-prescribed opioids or abuse of prescribed opioids.)
5. have a Karnofsky performance scale index score of >=60
6. provide informed consent
7. provide locator information
8. sign a HIPAA form / medical record release form to facilitate medical record abstraction
9. report living in the vicinity and being able to return for follow-up visits
10. complete the baseline assessment, including blood draw
11. be able to communicate in English

Exclusion Criteria

Individuals will be excluded from the study if they:

1. do not meet any one or more of the above-described inclusion criteria
2. have significant cognitive or developmental impairment to the extent that they are unable to provide informed consent
3. are terminated via Site PI decision with agreement from study Lead Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2012-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
HIV Viral Suppression | 12 months
  The primary outcome variable is binary: HIV viral suppression (<= 200 copies/ml), as determined by blood draw at/near the 12 month follow-up versus presence of viral load > 200 or death (all-cause mortality). We are aware that, for patients on therapy, the goal of antiretroviral therapy is achieving a viral load "below the limit of detection of the assay" which currently is usually < 40 copies/ml. However, we have chosen to define "suppression" as <= 200 copies/ml to be consistent with the January 2011 Guidelines for the Use of Antiretroviral Agents in HIV-1-Infected Adults and Adolescents.

SECONDARY OUTCOMES:
HIV Secondary Outcomes | 12 months
  1. Viral suppression at 6 months (binary; laboratory assay)
  2. CD4 Cell count (continuous; laboratory assay)
  3. Engagement into care (binary; self-report/medical record abstraction)
  4. HIV care visit attendance (count; self-report/medical record abstraction)
  5. Medication Adherence (count; self-report/ACTG Adherence Questionnaire)
  6. Hospitalizations (count; self-report/medical record abstraction)
  7. All cause mortality
Substance Use Related Secondary Outcomes | 12 months
  1. Substance use frequency (count; self-report ASI and binary; urine/breath analysis)
  2. Substance Use Severity (continuous, DAST and AUDIT)
  3. Treatment engagement (binary; self-report/medical record abstraction)
  4. Number of drug treatment sessions (Count; self-report/medical record abstraction)
Mediators and Moderators of Outcomes | 12 months
  1. Viral Suppression Moderators: psychological distress (BSI), Housing instability, Food Insecurity Health literacy, HIV-related cognitive problems, and renal and liver function status.
  2. Viral Suppression Mediators: Medication self-efficacy, Physician-Patient relationship, social support and substance use.
  3. CD4 Count Moderators: HCV status.
  4. Drug Use Moderators: Readiness for drug treatment
  5. Drug Use Mediators: Readiness for drug treatment and social support.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Metsch, Ph.D, Principal Investigator — Columbia University; Lauren Gooden, Ph.D, Study Director — Columbia University; Carlos del Rio, M.D., Principal Investigator — Emory University
Locations (12):
- United States (12):
  - University Hospital At University of Alabama, Birmingham (Uab), Birmingham, Alabama
  - Los Angeles County Harbor-UCLA Medical Center, Torrance, California
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami, Miami, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Stroger Cook County Hospital/Rush University Medical Center, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Saint Luke's Roosevelt Hospital Center, New York, New York
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (Upmc), Pittsburgh, Pennsylvania
  - Parkland Health and Human Services, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Information about the study and the de-identified study data will be available at https://datashare.nida.nih.gov/ within 18 months of the date the data are locked, as per the procedures of the National Drug Abuse Treatment Clinical Trials Network.

REFERENCES:
- [Derived] Gutkind S, Starbird LE, Murphy SM, Teixeira PA, Gooden LK, Matheson T, Feaster DJ, Jain MK, Masson CL, Perlman DC, Del Rio C, Metsch LR, Schackman BR. Cost of Hepatitis C care facilitation for HIV/Hepatitis C Co-infected people who use drugs. Drug Alcohol Depend. 2022 Mar 1;232:109265. doi: 10.1016/j.drugalcdep.2022.109265. Epub 2022 Jan 10. PMID 35042101
- [Derived] Stitzer ML, Gukasyan N, Matheson T, Sorensen JL, Feaster DJ, Duan R, Gooden L, Del Rio C, Metsch LR. Enhancing patient navigation with contingent financial incentives for substance use abatement in persons with HIV and substance use. Psychol Addict Behav. 2020 Feb;34(1):23-30. doi: 10.1037/adb0000504. Epub 2019 Aug 22. PMID 31436447
- [Derived] Mitchell SG, Monico LB, Stitzer M, Matheson T, Sorensen JL, Feaster DJ, Schwartz RP, Metsch L. How patient navigators view the use of financial incentives to influence study involvement, substance use, and HIV treatment. J Subst Abuse Treat. 2018 Nov;94:18-23. doi: 10.1016/j.jsat.2018.07.009. Epub 2018 Jul 22. PMID 30243412
- [Derived] Philbin MM, Feaster DJ, Gooden L, Duan R, Das M, Jacobs P, Lucas GM, Batey DS, Nijhawan A, Jacobson JM, Mandler R, Daar E, McMahon DK, Armstrong WS, Del Rio C, Metsch LR. The North-South Divide: Substance Use Risk, Care Engagement, and Viral Suppression Among Hospitalized Human Immunodeficiency Virus-Infected Patients in 11 US Cities. Clin Infect Dis. 2019 Jan 1;68(1):146-149. doi: 10.1093/cid/ciy506. PMID 29920584
- [Derived] Stitzer ML, Hammond AS, Matheson T, Sorensen JL, Feaster DJ, Duan R, Gooden L, Del Rio C, Metsch LR. Enhancing Patient Navigation with Contingent Incentives to Improve Healthcare Behaviors and Viral Load Suppression of Persons with HIV and Substance Use. AIDS Patient Care STDS. 2018 Jul;32(7):288-296. doi: 10.1089/apc.2018.0014. Epub 2018 Jun 8. PMID 29883190
- [Derived] Winhusen T, Feaster DJ, Duan R, Brown JL, Daar ES, Mandler R, Metsch LR. Baseline Cigarette Smoking Status as a Predictor of Virologic Suppression and CD4 Cell Count During One-Year Follow-Up in Substance Users with Uncontrolled HIV Infection. AIDS Behav. 2018 Jun;22(6):2026-2032. doi: 10.1007/s10461-017-1928-x. PMID 29030717
- [Derived] Stitzer M, Matheson T, Cunningham C, Sorensen JL, Feaster DJ, Gooden L, Hammond AS, Fitzsimons H, Metsch LR. Enhancing patient navigation to improve intervention session attendance and viral load suppression of persons with HIV and substance use: a secondary post hoc analysis of the Project HOPE study. Addict Sci Clin Pract. 2017 Jun 27;12(1):16. doi: 10.1186/s13722-017-0081-1. PMID 28651612
- [Derived] Metsch LR, Feaster DJ, Gooden L, Matheson T, Stitzer M, Das M, Jain MK, Rodriguez AE, Armstrong WS, Lucas GM, Nijhawan AE, Drainoni ML, Herrera P, Vergara-Rodriguez P, Jacobson JM, Mugavero MJ, Sullivan M, Daar ES, McMahon DK, Ferris DC, Lindblad R, VanVeldhuisen P, Oden N, Castellon PC, Tross S, Haynes LF, Douaihy A, Sorensen JL, Metzger DS, Mandler RN, Colfax GN, del Rio C. Effect of Patient Navigation With or Without Financial Incentives on Viral Suppression Among Hospitalized Patients With HIV Infection and Substance Use: A Randomized Clinical Trial. JAMA. 2016 Jul 12;316(2):156-70. doi: 10.1001/jama.2016.8914. PMID 27404184